CLINICAL TRIAL: NCT03882749
Title: A Multicenter Observational Study on the Use of Delivra-Celecoxib 8% Cream on Pain Experienced by Patients With Osteoarthritis of the Knees
Brief Title: Delivra-Celecoxib 8% Cream and Osteoarthritis
Acronym: Del-Cel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Delivra, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-OA-0001
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Pain, WOMAC
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The observation of the clinical use of the Delivra Celecoxib cream (8%) in the treatment of osteoarthritis of the knee. Observations will be made over 12 weeks of treatment. Evaluations include: pain, functionality and patients global assessment of disease. Patients will self administer treatment as prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients with primary osteoarthritis (with radiological evidence) of the knees who have been prescribed Del-Cel.
* On stable pain therapy with an oral or topical NSAID or acetaminophen.
* Able to read and understand English to answer pain assessment questions independently.
* Willing and able to fulfill the requirements of the study, including complete scheduled follow-up phone visits.

Exclusion Criteria:

* Inability to adequately read and understand English as required to complete study assessments and comply with the protocol.
* Current recreational or medicinal use of cannabis within 4 weeks of study initiation.
* Participants with a lifetime history of cannabis use disorder or other substance use disorders (except tobacco use disorder) will be excluded.
* Participants with a lifetime history of daily cannabis use will be excluded.
* Dose changes of concomitant medication will not be permitted during the study period.
* Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months), or women who are planning on becoming pregnant.
* Diagnosis of any of the following mental disorders as defined by the DSM-5: a lifetime history of schizophrenia or any other psychosis, organic medical disorders, bipolar disorder. Entry of patients with obsessive compulsive disorder or post- traumatic stress disorder will be permitted if the anxiety disorder is judged to be the predominant disorder, in order to increase accrual of a clinically relevant sample.
* Major depression will be allowed if not severe (Montgomery Åsberg Depression Rating Scale-MADRS27≥ 25). Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
* Participants with a family history of schizophrenia spectrum or bipolar disorder will be excluded.
* Participants who have a history of adverse reactions to cannabis will be excluded.
* Known allergy to any of the ingredients in the Delivra base.
* Use of Rimonabant (SR141716) within three weeks of enrollment and/or planned use for the duration of the study participation[27].
* Use of 5-HT1A receptor antagonists (SSRI inhibitors) within three weeks of enrollment and/or planned use for the duration of the study participation, e.g.: Pindolol, Lecozotan, Brexpiprazole, etc.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population is all patients prescribed Del-Cel for the treatment of Osteoarthritis of the knees. The treating rheumatologist/ attending clinician will determine the appropriate course of treatment for patients as per routine clinical practice. Only patients prescribed Del-Cel will be approached for informed consent and voluntary participation in this observational study.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-07-23 (Estimated); Study Completion 2019-10-23 (Estimated)

PRIMARY OUTCOMES:
11-Point Numerical Rating Scale Pain Index | over 12 weeks
  Subjects will rate he pain that they experience from 0-no pain to 10-worst pain inmmaginable
WOMAC | over 12 weeks
  Subjects will describe pain and functionality status using a validated likert assessment .

SECONDARY OUTCOMES:
Adverse event reporting | over 12 weeks
  Subjects will report any adverse events experienced during the study

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Dr. Angela Montgomery - Rheumatologist, Mississauga, Ontario
  - Dr. Brandusa Florica - Rheumatologist, Mississauga, Ontario
  - Dr. Andrew Chow - Rheumatologist, Mississauga, Ontario